CLINICAL TRIAL: NCT04224454
Title: Influenza, Pneumococcal and Diphtheria-tetanus-poliomyelitis Vaccine Coverage in Patients With Primary Sjögren's Syndrome: a Cross-sectional Study
Brief Title: Vaccine Coverage and Primary Sjögren'Syndrome
Acronym: VACGREN
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0612
Record Dates: First submitted 2020-01-02; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Primary Sjögren Syndrome
Keywords: Vaccine; Coverage; Sjögren's syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary Sjögren's syndrome: 111 consecutive patients with primary Sjögren's syndrome (European-American 2002 criteria)
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire was adapted from questionnaires used by the French national agency "Institut de Veille Sanitaire" to study vaccination coverage and were completed with the assistance of one fellow to limit missing data.

SUMMARY:
Evaluation of vaccination coverage for influenza, pneumococcus and DTP in patients with pSS and investigated the reasons for non-vaccination.

DETAILED DESCRIPTION:
A cross-sectional study was performed in pSS patients from two different French tertiary referral centers for autoimmune diseases (Paris-Bicêtre and Montpellier). From January 2016 to November 2017, questionnaires were randomly delivered to patients with pSS according to European-American Diagnostic Criteria (2002). Before completing the questionnaire, patients gave their consent to participate. This questionnaire was adapted from questionnaires used by the French national agency "Institut de Veille Sanitaire" to study vaccination coverage and were completed with the assistance of one fellow (HL) to limit missing data.

Data collected in the questionnaire included previous vaccinations, reasons for non-vaccination, sources of vaccine proposition, and sociodemographic data including education level (Bachelor degree, and post-Bachelor degree education) and presence of young child(ren) (inferior 10 years old) at home. The following data was collected from the medical file: European-American Diagnostic Criteria (2002) for pSS, the most recent EULAR Sjögren's syndrome disease activity index (ESSDAI), comorbidities (chronic lung diseases, diabetes, chronic kidney diseases, chronic liver diseases, chronic heart diseases, cardiovascular comorbidities [coronary or cerebral ischemia] and severe neurological or muscle diseases), history of severe A cross-sectional study was performed in pSS patients from two different French tertiary referral centers for autoimmune diseases (Paris-Bicêtre and Montpellier). From January 2016 to November 2017, questionnaires were randomly delivered to patients with pSS according to European-American Diagnostic Criteria (2002). Before completing the questionnaire, patients gave their consent to participate. This questionnaire was adapted from questionnaires used by the French national agency "Institut de Veille Sanitaire" to study vaccination coverage and were completed with the assistance of one fellow (HL) to limit missing data. Data collected in the questionnaire included previous vaccinations, reasons for non-vaccination, sources of vaccine proposition, and sociodemographic data including education level (Bachelor degree, and post-Bachelor degree education) and presence of young child(ren) (inferior 10 years old) at home. The following data was collected from the medical file: European-American Diagnostic Criteria (2002) for pSS, the most recent EULAR Sjögren's syndrome disease activity index (ESSDAI), comorbidities (chronic lung diseases, diabetes, chronic kidney diseases, chronic liver diseases, chronic heart diseases, cardiovascular comorbidities [coronary or cerebral ischemia] and severe neurological or muscle diseases), history of severe infection (requiring intravenous antibiotics or hospital admission), current smoking status, treatments used for pSS including hydroxychloroquine, immunosuppressive drugs (methotrexate, leflunomide, ciclosporine, azathioprine, mycophenolate mofetil) and biological disease-modifying anti-rheumatic drugs (bDMARDs).

For descriptive statistical analysis, mean more or less SD were used for continuous variables and frequencies (percentage) for categorical variables. To evaluate factors associated with up-to-date vaccination, the investigators compared categorical variables between patients with updated and non-updated influenza, pneumococcal or DTP vaccines by using the Fisher exact test or chi-square test as appropriate. Continuous variables (age, ESSDAI) were compared by Student t test. A binary logistic regression model was used for multivariate analysis to estimate the odds ratio (OR) of being vaccinated with the 95% confidence interval (CI). p< 0.05 was considered statistically significant. All statistical analyses were performed with IBM SPSS 15 software.

ELIGIBILITY:
Inclusion criteria:

- patients with pSS according to European-American Diagnostic Criteria

Exclusion criteria:

- Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with primary Sjögren'syndrome
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of patients with Sjögren's syndrome vaccinated against influenzae virus | 1 year
  Rate of patients with Sjögren's syndrome vaccinated against influenzae virus: number of patients vaccinated against influenzae virus within 1 year divided to the number of patients not vaccinated against influenzae virus within 1 year
Rate of patients with Sjögren's syndrome vaccinated against streptococcus pneumoniae | 5 years
  Rate of patients with Sjögren's syndrome vaccinated against streptococcus pneumoniae: number of patients vaccinated against streptococcus pneumoniae within 5 years divided to the number of patients not vaccinated against streptococcus pneumoniae within 5 years
Rate of patients with Sjögren's syndrome vaccinated against DTP | 10 years
  Rate of patients with Sjögren's syndrome vaccinated against DTP : number of patients vaccinated for DTP within 10 years divided to the number of patients not vaccinated for DTP within 10 years

SECONDARY OUTCOMES:
Evaluate the reasons for non-vaccination | 1 day
  Evaluate the reasons for non-vaccination : The questionnaire was adapted from questionnaires used by the French national agency "Institut de Veille Sanitaire" to study vaccination coverage and were completed with the assistance of one fellow (HL) to limit missing data (18). Data collected in the questionnaire included previous vaccinations, reasons for non-vaccination, sources of vaccine proposition, and sociodemographic data including education level (Bachelor degree, and post-Bachelor degree education) and presence of young child(ren) (<10 years old) at home.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques MOREL, Professor, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Background] Gluthmann J FL, Bonmarin I, Levy-Bruhl D. Enquête nationale de couverture vaccinale, France, janvier 2011. http://www.invs.sante.fr. . 2001.